CLINICAL TRIAL: NCT00227305
Title: A 26-week, Multicenter, Open-label Phase 3b Study of the Safety and Tolerability of Quetiapine Fumarate (SEROQUEL™) Immediate-release Tablets in Daily Doses of 400 mg to 800 mg in Children and Adolescents With Bipolar I Disorder and Adolescents With Schizophrenia (Abbreviated)
Brief Title: Quetiapine Fumarate (SEROQUEL) in the Treatment of Adolescent Patients With Schizophrenia and Bipolar I Disorder
Acronym: ANCHOR 150
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1441C00150
Record Dates: First submitted 2005-09-27; First posted 2005-09-28 (Estimated); Results first posted 2012-10-05 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia; Bipolar I Disorder
Keywords: Schizophrenia; Bipolar I Disorder
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: quetiapine fumarate — Oral dosing, flexible dosing
  Other Names: Seroquel

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of quetiapine fumarate (SEROQUEL) in the treatment of adolescent patients with schizophrenia and bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to provide written assent and the parents or legal guardian of the patient are/is able to provide written informed consent before beginning any study related procedures
* Patient previously enrolled in either double-blind Study D1441C00149 or D1441C00112
* Patient has documented clinical diagnosis of schizophrenia or bipolar I disorder
* Patient's parent or legal guardian will be able to accompany the patient to each scheduled study visit

Exclusion Criteria:

* Patients (female) must not be pregnant or lactating
* Patients with a known intolerance or lack of response to previous treatment with quetiapine
* Patients who have previously participated in this study

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 381 (Actual)
Dates: Start 2004-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (48):
- United States (31):
  - Research Site, Dothan, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Cerritos, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Denver, Colorado
  - Research Site, Altamonte Springs, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Oak Brook, Illinois
  - Research Site, Newton, Kansas
  - Research Site, Overland Park, Kansas
  - Research Site, New Orleans, Louisiana
  - Research Site, Las Vegas, Nevada
  - Research Site, Rochester, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Lyndhurst, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Kirkland, Washington
  - Research Site, Milwaukee, Wisconsin
- Research Site, Lucknow, India
- Malaysia (2):
  - Research Site, Kuala Lumpur
  - Research Site, Petaling Jaya
- Philippines (4):
  - Research Site, Davao City
  - Research Site, Mandaluyong
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (2):
  - Research Site, Poznan
  - Research Site, Torun
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Novi Sad
- Research Site, Pretoria, South Africa
- Ukraine (3):
  - Research Site, Kharkiv
  - Research Site, Lviv
  - Research Site, Odesa

REFERENCES:
- [Derived] Findling RL, Pathak S, Earley WR, Liu S, DelBello M. Safety, tolerability, and efficacy of quetiapine in youth with schizophrenia or bipolar I disorder: a 26-week, open-label, continuation study. J Child Adolesc Psychopharmacol. 2013 Sep;23(7):490-501. doi: 10.1089/cap.2012.0092. Epub 2013 Sep 11. PMID 24024534

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was contingent on completing one of 2 short term efficacy studies, recruitment period August 2004 through July 2007 at 59 international clinical research sites
Pre-assignment Details: Required to have completed one feeder study, either bipolar mania study D1441C00149 or schizophrenia study D1441C00112 and be willing to participate in a 26 week open label study and be between the ages of 10 and 18 years at the time of consent for this study, initial titration to maintain blind in feeder study
Groups:
- Quetiapine: Quetiapine 400mg/day to 800mg/day
Period: Overall Study
Arm/Group | Quetiapine
Started | 381 (enrolled)
Drug Received | 380 (safety population)
Completed | 237 (Completed 26 weeks)
Not Completed | 144
Not completed — Adverse Event | 40
Not completed — Withdrawal by Subject | 42
Not completed — Lost to Follow-up | 33
Not completed — Study specific discontinuation | 13
Not completed — MOVED OUT OF AREA | 3
Not completed — Lack of Efficacy | 7
Not completed — Physician Decision | 3
Not completed — PERIOD SHORTENED FROM 6 wks to 4 wks | 1
Not completed — LEAVING TOWN FOR 6 WEEKS | 1
Not completed — NECESSITY OF USING ANTI DEPRESSANT | 1

BASELINE CHARACTERISTICS:
Arm/Group | Quetiapine
Number analyzed (Participants) | 380
Age, Customized [Number; unit: Participants]
  10 - 12 years | 87
  13 - 18 years | 293
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154
  Male | 226
Diagnosis [Number; unit: participant from feeder studies]
  Bipolar | 205
  Schizophrenia | 175

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Nature of Adverse Events (AEs)
Description: Number of participants that had AE which occurred from first dose date to last dose date + 30 days.
Time Frame: from open label to week 26+ 30 days
Measure: Number; unit: Participants
Arm/Group | Quetiapine
Number analyzed (Participants) | 380
Participants | 321

2. Primary Outcome: Number of Patients Withdrawn Due to AEs.
Description: Number of subjects who withdrew from the study due to AEs.
Time Frame: during 26 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Quetiapine
Number analyzed (Participants) | 380
Participants | 37

3. Primary Outcome: Changes in Laboratory Test Results (Prolactin)
Description: Clinical important shift to high prolactin from open-label (OL) baseline to week 26.
  High Prolactin is defined as value >26 ug/L for female and value >20 ug/L for male.
Time Frame: Duration of study participation
Measure: Number; unit: Participants
Arm/Group | Quetiapine
Number analyzed (Participants) | 380
Participants | 19

4. Secondary Outcome: Changes in Tanner Stage
Description: Category shift in Tanner stage. Number of subjects who experienced the change is presented.
  Tanner stages (I-V) was used to characterize physical development in children, adolescents, and adults. The stages was based on external primary and secondary sex characteristics, such as the size of the breasts, genitalia, and development of pubic hair. Tanner stage is considered going up when the organs grow bigger.
Time Frame: Change from OL baseline to week 26 in the Tanner stage
Population: Number of patients with Tanner stagging data at OL baseline and week 26 (final visit)
Measure: Number; unit: Participants
Arm/Group | Quetiapine
Number analyzed (Participants) | 373
Participants | 70

5. Secondary Outcome: Change From Baseline in Children's Global Assessment Scale (CGAS) Score
Description: Children's Global Assessment Scale (CGAS) is used to rate the general functioning of children under the age of 18. It is the 100-point single-item score that was collected in the Clinical Report Form (CRF), scored from 0-100 (worse to normal).
Time Frame: OL Baseline to Week 26
Population: Number of patients with CGAS score at OL baseline and week 26.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine
Number analyzed (Participants) | 320
units on a scale | 7 (13.9)

6. Primary Outcome: Categorical Change From OL Baseline to Week 26 in Simpson-Angus Scale (SAS)Total Score
Description: Number of patients for who the total score is estimated as worse. The Simpson Angus Scale (SAS)is used to assess Parkinsonian symptoms (a type of movement disorders). The score was calculated as the sum of the 10 individual item scores. Total Score ranges from 0-40 (normal to worse). Individual item scale range from 0 to 4 (normal to worse).
  Improved define as those with a <= -1 change in SAS total score. Worsened defined as those with a >=1 change in SAS total score.
Time Frame: OL baseline to week 26
Population: Number of patients with SAS score at OL baseline and week 26.
Measure: Number; unit: Participants
Arm/Group | Quetiapine
Number analyzed (Participants) | 373
Participants | 34

7. Primary Outcome: Categorical Change From Baseline in Barnes Akathisia Rating Scale (BARS) Global Score
Description: Number of patients for who the total score is estimated as worse. The Barnes Akathisia Rating Scale (BARS) global score is used to measure Akathisia (a type of movement disorders). BARS is the item 4 score from the BARS assessment. The scale is from a range 0-5 (normal to worse). Change from baseline in BARS global score increase means worse.
  Improved defined as those with a <= -1 change in BARS global score. Worsened defined as those with a >= 1 change in BARS global score.
Time Frame: 26 weeks of treatment
Population: Number of patients with BARS score at OL baseline and week 26.
Measure: Number; unit: Participants
Arm/Group | Quetiapine
Number analyzed (Participants) | 373
Participants | 11

8. Primary Outcome: Change From Baseline in Weight
Description: Number with 7% or more increase (without adjustment for normal growth)
Time Frame: 26 weeks of treatment
Population: Number of participants is based on patients with both baseline values and post-baseline values.
Measure: Number; unit: Participants
Arm/Group | Quetiapine
Number analyzed (Participants) | 373
Participants | 134

9. Primary Outcome: Change From Baseline in Supine Pulse
Description: Change from OL baseline to week 26 in supine pulse (bpm)
Time Frame: OL baseline to week 26
Population: Number of participants with OL baseline and post treatment visits
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Quetiapine
Number analyzed (Participants) | 375
bpm | 0.8 (14.75)

10. Primary Outcome: Change From OL Baseline in Supine Systolic BP.
Description: Changes from OL baseline to the final visits in Supine systolic BP (mmHg)
Time Frame: OL baseline to Week 26
Population: Number of participants with OL baseline and post treatment visits
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Quetiapine
Number analyzed (Participants) | 375
mmHg | 1.7 (11.52)

11. Primary Outcome: Change From OL Baseline in Supine Diastolic BP.
Description: Changes from OL baseline to the final visits in Supine diastolic BP (mmHg)
Time Frame: OL baseline to Week 26
Population: Number of participants with OL baseline and post treatment visits
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Quetiapine
Number analyzed (Participants) | 375
mmHg | 1.3 (9.22)

ADVERSE EVENTS:
Time Frame: Other AE module includes adverse events which occurred before first dose date to last dose date + 30 days.
Arm/Group | Quetiapine
Serious Adverse Events (participants affected / at risk) | 46/380
Other Adverse Events (participants affected / at risk) | 340/380
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine (N=380)
Abnormal Behaviour (Psychiatric disorders) | 1
Aggression (Psychiatric disorders) | 4
Agitation (Psychiatric disorders) | 1
Amoebiasis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 2
Bacterial Infection (Infections and infestations) | 1
Bipola Disorder (Psychiatric disorders) | 12
Cellulitis Staphylococcal (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1
Delusion (Psychiatric disorders) | 1
Disinhibition (Psychiatric disorders) | 1
Drug Toxicity (Injury, poisoning and procedural complications) | 1
Hallucitnation Auditory (Psychiatric disorders) | 1
Hostility (Psychiatric disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypertensive Crisis (Vascular disorders) | 1
Irritability (General disorders) | 1
Mania (Psychiatric disorders) | 1
Myocarditis Post Infection (Cardiac disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Overdose (Injury, poisoning and procedural complications) | 2
Perceptual Alteration Paroxysmal (Psychiatric disorders) | 1
Physical Assault (Vascular disorders) | 1
Pyschotic Disorder (Psychiatric disorders) | 2
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pyrexia (Respiratory, thoracic and mediastinal disorders) | 1
Restlessness (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 8
Schizophrenia, Paraniod Type (Psychiatric disorders) | 1
Staphylococcal Infection (Infections and infestations) | 1
Suicide Attempt (Psychiatric disorders) | 1
Syncope (Nervous system disorders) | 1
Typhoid Fever (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine (N=380)
AGITATION (Psychiatric disorders) | 26
DIZZINESS (Nervous system disorders) | 26
DRY MOUTH (Gastrointestinal disorders) | 35
FATIGUE (Gastrointestinal disorders) | 20
HEADACHE (Nervous system disorders) | 43
INCREASED APPETITE (Metabolism and nutrition disorders) | 76
INSOMNIA (Psychiatric disorders) | 43
IRRITABILITY (Psychiatric disorders) | 23
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 20
NAUSEA (Gastrointestinal disorders) | 39
SEDATION (Nervous system disorders) | 72
SOMNOLENCE (Nervous system disorders) | 115
TACHYCARDIA (Cardiac disorders) | 25
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 27
VOMITING (Gastrointestinal disorders) | 43
WEIGHT INCREASED (Gastrointestinal disorders) | 65

LIMITATIONS AND CAVEATS:
No comparator group, open label treatment, duration only 26 weeks - not long enough to assess full impact on growth and development

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca as sponsor will first publish results for the multicenter study